CLINICAL TRIAL: NCT06418568
Title: Efficacy and Safety Trial of Using Ultra-Pulsed Shockwaves to Deliver Tranexamic Acid for the Treatment of Melasma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1174
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Chloasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with chloasma (Experimental): The intervention involves treating melasma using tranexamic acid (aminomethylbenzoic acid) delivered through ultra-pulsed shockwave therapy on one side of the face, while the other side receives topical application of tranexamic acid at the same concentration.
  Interventions: Device: Ultra-pulsed Shockwave Therapy Device by Shenzhen Lifotronic Technology Co., Ltd.

INTERVENTIONS:
Device: Ultra-pulsed Shockwave Therapy Device by Shenzhen Lifotronic Technology Co., Ltd. — The intervention involves treating melasma using tranexamic acid (aminomethylbenzoic acid) delivered through ultra-pulsed shockwave therapy on one side of the face, while the other side receives topical application of tranexamic acid at the same concentration. The shockwave therapy parameters are tailored based on patient tolerance. Each patient undergoes 3 treatment sessions spaced 3 weeks apart, followed by a 4-week follow-up period. Facial skin is assessed using the VISIA system before each treatment and at the 4-week follow-up, evaluating the Melasma Area Severity Index (MASI). Patient and researcher satisfaction levels are rated on a scale of 1 to 5. Adverse reactions, including short-term effects like pain and swelling, and potential long-term effects such as allergic reactions and hyperpigmentation, are monitored after each treatment session.

SUMMARY:
Melasma is a prevalent chronic facial pigmentation condition affecting Asian women of childbearing age, attributed to genetic predisposition, sunlight exposure, and hormonal changes. Treatment methods include phototherapy and medication, notably tranexamic acid, which inhibits melanin production. Ultra-pulsed shockwave therapy is a non-invasive approach that boosts skin cell vitality and collagen synthesis.

Currently, there is a lack of comprehensive research on the effectiveness and safety of using ultra-pulsed shockwaves to deliver tranexamic acid for melasma treatment. This study will involve a non-randomized, self-half-face, pre-post controlled prospective clinical trial. This design aims to evaluate the depigmenting effects and safety profile of tranexamic acid delivered via ultra-pulsed shockwaves.

DETAILED DESCRIPTION:
Melasma is a common, chronic, acquired facial pigmentation disorder, also known as chloasma. Clinically, it presents as symmetrical, unevenly pigmented light to dark brown patches on the cheeks, forehead, and jawline with indistinct borders. The prevalence among Asian women of childbearing age can be as high as 30%, and it tends to recur and is difficult to cure.

The pathogenesis of melasma is not fully understood, but genetic susceptibility, sunlight exposure, and hormonal changes are considered the three major contributing factors. Increased melanin synthesis, vascular proliferation at skin lesions, inflammation, and impaired skin barrier all play roles in the development of melasma.

Melasma is clinically staged as active or stable phase. Clinical subtypes of melasma are categorized based on vascular involvement into 2 types: pure pigment type (M-type) and pigment combined with vascular type (M + V type). This classification guides the selection of treatment drugs and methods. According to the location of pigmentation, it is classified into 2 types: epidermal type (increased epidermal pigmentation) and mixed type (increased epidermal pigmentation + dermal superficial melanocytes). This classification is useful for determining treatment efficacy.

In the Expert Consensus on Phototherapy and Repair of Melasma (2020 edition), it is suggested that systemic medication is not the first choice for treating melasma and is mostly used off-label. Intravenous administration is effective, and oral administration is generally less effective. Common regimens include vitamin C, glutathione combined with vitamin C, and intravenous tranexamic acid. Oral tranexamic acid has some efficacy.

The Expert Consensus on the Diagnosis and Treatment of Melasma in China (2021 edition) states that single or repeated phototherapy can lead to pigment deposition, pigment reduction/loss, and recurrence, thus phototherapy is not recommended as a long-term clinical maintenance approach. The number of consecutive phototherapy treatments should not exceed 15 times, and repeat treatments can be considered after a 1-year interval. Topical medication is the preferred treatment: 1. Photoprotective agents, routinely combined with antioxidants; 2. Hydroquinone and its combination therapy are the most thoroughly researched topical medications. Adverse reactions include skin irritation, allergic contact dermatitis, and rarely, ochronosis; 3. Non-hydroquinone topical medications: retinoic acid, tranexamic acid, kojic acid, mequinol, arbutin, licorice extract, niacinamide, etc., most of which are also tyrosinase inhibitors.

Tranexamic acid, also known as aminomethylbenzoic acid, is clinically used primarily for various bleeding disorders caused by acute or chronic, localized, or systemic primary fibrinolysis. Tranexamic acid is a protease inhibitor, with a molecular structure very close to tyrosine. When high concentrations of tranexamic acid enter skin tissues, it competitively binds with tyrosinase, inhibiting its activity and thereby reducing melanin formation. Therefore, tranexamic acid has been widely used clinically in dermatology for the treatment of melasma both domestically and abroad.

Tranexamic acid's main indication in clinical practice is hemostasis. Oral tranexamic acid for treating melasma is considered off-label, and long-term oral administration carries risks such as thrombosis (cerebral thrombosis, myocardial infarction, venous thrombosis, etc.), necessitating long-term monitoring of patients' coagulation function and blood viscosity. Therefore, topical application of tranexamic acid directly to the affected skin area can enhance local drug efficacy and significantly reduce systemic adverse reactions due to its effect on the skin barrier; however, the local effective absorption rate of topically applied tranexamic acid is the main limitation for achieving therapeutic effects.

Ultra-pulsed shockwave therapy is a non-invasive anti-aging treatment that can be applied to facial rejuvenation. It uses the principle of high-speed vibration to compress the medium intensely and focus to generate mechanical sound waves. Mechanical sound waves produce physical effects on the skin, including mechanical effects, shockwave technical effects, and cavitation effects, to activate biological effects, among which a 36mm treatment handle acts on superficial tissues, improving local cell membrane permeability and can be used for drug-related delivery, enhancing cellular vitality and metabolic capacity, stimulating collagen regeneration.

Tranexamic acid delivery therapy is a common treatment method for melasma, while utilizing ultra-pulsed shockwaves to deliver tranexamic acid is a novel treatment approach. Currently, there is no comparative research on the efficacy and safety of tranexamic acid (aminomethylbenzoic acid) delivered via ultra-pulsed shockwave therapy for treating melasma domestically and internationally. This study designs a non-randomized, self-half-face, and pre-post controlled prospective clinical trial, intending to use ultra-pulsed shockwaves to deliver tranexamic acid to increase local tranexamic acid concentration in the skin spots and achieve depigmenting effects safely. This will provide clinical evidence for dermatologists and patients to formulate individualized treatment plans.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, any gender;
2. Diagnosis of melasma;
3. Able to comprehend and voluntarily sign a written informed consent form, and able to complete the treatment and follow-up as required.

Exclusion Criteria:

1. History of other pigmentary disorders such as lentigines, Ota nevus, freckles, etc.;
2. History of oral retinoid or tetracycline-class photosensitizing drugs within the past 6 months prior to treatment;
3. History of facial injections, fillers, chemical peels, laser or radiofrequency treatments, or other treatments targeting pigmentation within the past 6 months prior to treatment;
4. Abnormal coagulation function;
5. History of oral glucocorticoids or immunosuppressive agents within the past 3 months prior to treatment;
6. Patients with malignant tumors;
7. Pregnant or lactating women;
8. Patients with active herpes simplex or herpes zoster on the face.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Melasma area severity index(MASI) | 3 months
  The Melasma Area Severity Index (MASI) is a clinical scoring system used to assess the severity of melasma based on the extent and darkness of pigmented areas on the face. It takes into account four different facial regions: the forehead, cheeks (right and left), and chin.
  The MASI score is calculated using the following formula:
  MASI=0.3×(DF+DB)×AF+0.3×(RF+RB)×AF+0.3×(CF+CB)×AF+0.1×(LF+LB)×AF
  The MASI score ranges from 0 to approximately 48, with higher scores indicating more severe melasma. It is used to quantify and monitor changes in melasma severity over time in response to treatment interventions.

SECONDARY OUTCOMES:
Physician's Global Assessment (PGA) | 3 months
  Physician's Global Assessment (PGA) Overall Evaluation by Physicians: Based on the residual condition of pigmentation after treatment, scores range from 0 to 6 points:
  0 points indicate complete clearance (100%) or minimal residual pigmentation,
  1. point indicates essentially cleared (≥ 90%),
  2. points indicate marked improvement (75% ~ 89%),
  3. points indicate moderate improvement (50% ~ 74%),
  4. points indicate slight improvement (25% ~ 49%),
  5. points indicate no improvement (< 25%),
  6. points indicate worsening compared to before treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China